CLINICAL TRIAL: NCT04582253
Title: Pix2pix Conditional Generative Adversarial Networks for Scheimpflug Camera Color-coded Corneal Tomography Image Generation
Brief Title: Pix2pix Networks for Scheimpflug Corneal Tomography Image Generation
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Abdelazeem, Associate professor of Ophthalmology, Assiut University
Other Study IDs: 17300483
Record Dates: First submitted 2020-10-05; First posted 2020-10-09 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Eye Diseases
Keywords: Cornea; Imaging
MeSH Terms: conditions — Eye Diseases; Corneal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Keratoconus: Those with a clinical diagnosis of keratoconus such as:
  a) the presence of a central protrusion of the cornea with Fleischer ring, Vogt striae, or both by slitlamp examination.(b) an irregular cornea determined by distorted keratometry mires and distortion of retinoscopic red reflex or both in addition to the following topographic findings as summarized by Pińero and colleagues: focal steepening located in a zone of protrusion surrounded by concentrically decreasing power zones, focal areas with dioptric (D) values >47.0D, inferior- superior(I-S) asymmetry measured to be > 1.4 D or angling of the hemimeridians in an asymmetric or broken bowtie pattern with skewing of the steepest radial axis (SRAX) 2.
  Interventions: Diagnostic Test: Scheimpflug Camera Corneal Tomography
- Subclinical keratoconus: Defined as subtle corneal tomographic changes as the aforementioned keratoconus abnormalities in the absence of slit- lamp or visual acuity changes typical of keratoconus (subclinical keratoconus).
  Interventions: Diagnostic Test: Scheimpflug Camera Corneal Tomography
- Normal: This group comprised refractive surgery candidates and subjects applying for a contact lens fitting with a refractive error of less than 8.0 D sphere with less than 3.0 D of astigmatism and without clinical, topographic or tomographic signs of keratoconus nor suspected keratoconus.
  Interventions: Diagnostic Test: Scheimpflug Camera Corneal Tomography

INTERVENTIONS:
Diagnostic Test: Scheimpflug Camera Corneal Tomography — Pentacam Sheimpflug system(Pentacam HR, Oculus Optikgeräte GmbH, software V.1.15r4 n7) is used for imaging of the anterior and posterior surfaces of the cornea to obtain corneal tomographic maps.

SUMMARY:
Computer-aided medical image analysis has advantages, but requires large amounts of training data, which are scarce and costly to obtain, are subject to privacy concerns, and are often highly imbalanced, with over-representation of common conditions and poor representation of rare conditions. Consequently, some methods have been proposed to generate artificial medical images using generative adversarial networks (GANs). Computer aided diagnosis of keratoconus is an emerging research field that may benefit greatly from medical image synthesis, which can affordably provide an arbitrary number of sufficiently diverse synthetic images that mimic real Pentacam images. A new conditional GAN, the pix2pix cGAN, has not been used in this context to date. Here, investigators will assess the efficacy of a cGAN implementing pix2pix image translation for image synthesis of color-coded Pentacam 4-map refractive displays of clinical and subclinical keratoconus as well as normal corneas.

ELIGIBILITY:
Inclusion Criteria:

* Keratoconus group:

  * Presence of a central protrusion of the cornea with Fleischer ring, Vogt striae, or both by slitlamp examination.
  * irregular cornea determined by distorted keratometry mires and distortion of retinoscopic red reflex or both in addition to the following topographic findings as summarized by Pińero and colleagues :
  * focal steepening located in a zone of protrusion surrounded by concentrically decreasing power zones
  * focal areas with dioptric (D) values >47.0D
  * inferior- superior(I-S) asymmetry measured to be > 1.4 D
  * Angling of the hemimeridians in an asymmetric or broken bowtie pattern with skewing of the steepest radial axis(SRAX) .

Suspicious group:

• Defined as subtle corneal tomographic changes as the aforementioned keratoconus abnormalities in the absence of slit- lamp or visual acuity changes typical of keratoconus (forme fruste keratoconus).

Normal group:

* Refractive surgery candidates
* Refractive error of less than 8.0 D sphere
* Less than 3.0 D of astigmatism
* without clinical, topographic or tomographic signs of keratoconus or suspect keratoconus.

Exclusion Criteria:

* • Systemic disease

  * Other corneal disease such as pellucid marginal degeneration
  * History of trauma
  * Corneal surgery such as corneal cross- linking for progressive keratoconus.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Refractive surgery candidates with unilateral, bilateral, or forme fruste keratoconus, obtained between July 2014 and March 2019 at private eye center, Assiut, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 923 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Scheimpflug camera color-coded corneal tomography images created by pix2pix conditional adversarial network (pix2pix cGAN) | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No